CLINICAL TRIAL: NCT03648398
Title: Pilot Study of an Online Therapeutic Education Program for Patients With Inflammatory Bowel Disease
Acronym: EDUMICILOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Muriel VELTIN, Nurse, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APPARA2018/EDUMICILOR-VELTIN
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Therapeutic education program; Online
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EDUMICILOR (Other): Patients will participate in the online therapeutic education program for about 6 months
  Interventions: Other: EDUMICILOR

INTERVENTIONS:
Other: EDUMICILOR — Patients will participate in the online therapeutic education program for about 6 months

SUMMARY:
EDUMICILOR is a monocentric prospective pilot study for patients with inflammatory bowel disease (IBD).

During the study, patients will participate in an online therapeutic education program.

They will first have an appointment with a nurse to establish a personalized educational diagnosis. Then they will participate in the online therapeutic education program for about 6 months (depends on the educational needs, expectations and patient's availabilities).

The main objective of this study is to assess the feasibility of an online therapeutic education program for IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (age ≥ 18 years old)
* Patients with established Crohn's disease or ulcerative colitis diagnosis
* Patients who own the equipment to participate in the online therapeutic education program (computer, webcam….)
* French speaking patients
* Patients who cannot attend regular therapeutic education sessions at the hospital
* Patients able to understand the information provided to them and to give written informed consent for the study

Exclusion Criteria:

* Patient who has not given his/her consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of participation in the online therapeutic education program | 6 months
  Patients must participate in at least 80% of therapeutic education program sessions and connect to at least one video or one serious game.

SECONDARY OUTCOMES:
Score of the Crohn and Colitis Knowledge Score | 6 months
  The Crohn and Colitis Knowledge Score will assess the impact of the online therapeutic education program on achieving educational objectives.
Score of the short Inflammatory Bowel Disease Questionnaire (short-IBDQ) | 6 months
  The short-IBDQ will assess the quality of life before and after the online therapeutic education program.
Score of the Inflammatory Bowel Disease Disability Index (IBD Disability Index) | 6 months
  The IBD Disability index will be used to assess disability before and after the online therapeutic education program.
Score of the Hospital Anxiety and Depression Scale | 6 months
  The Hospital Anxiety and Depression scale will assess the anxiety and depression level before and after the online therapeutic education program.
Score of the Girerd Scale | 6 months
  The Girerd Scale will be used to assess the level of adherence to prescribed drugs before and after the online therapeutic education program.
Score of a satisfaction survey on the online therapeutic education program | 6 months
  This survey will identify the advantages and disadvantages of an online therapeutic education program.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Veltin, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- CHRU Nancy, Nancy, France